CLINICAL TRIAL: NCT05815355
Title: Efficacy of Exclusive Enteral Nutrition in Adult Active Crohn's Disease With Complications or Failure of Medical Treatment
Brief Title: Efficacy of Exclusive Enteral Nutrition in Adult Active Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiang Peng, Attending physician, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: E2016008
Record Dates: First submitted 2022-09-25; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

INTERVENTIONS:
Dietary Supplement: exclusive enteral nutrition treatment group

SUMMARY:
Patients with Crohn's disease (CD) could develop complications such as stricture, intestinal fistula and abdominal abscess. Some CD patients had poor response to medical therapy. The efficacy of exclusive enteral nutrition (EEN) to these adult active CD patients is still unclear. The investigators aim to study the efficacy of EEN in induction of remission in adult active CD patients with complications or poor response to drugs.

DETAILED DESCRIPTION:
Active CD patients following up in our center who had been diagnosed as complicated disease with stricture, intestinal fistula, abdominal abscess and no response to drugs, were recruited since July 2013. Patients were only offered EEN for 12 weeks without using other drugs except that patients with abscess could use antibiotic therapy with or without percutaneous drainage. The disease activity was assessed by the Crohn's disease activity index (CDAI). CDAI<150 was taken as achieving clinical remission. Demographics and clinical variables were recorded. Nutritional (body mass index, albumin) and inflammatory (High sensitivity C-reactive protein and platelet) index were evaluated at baseline, week 4 and week 12. Some patients performed colonoscopy and/or computed tomography enterography (CTE) /resonance enterography(MRE) before and after EEN. Mucosal healing was assessed under endoscopy with SES-CD and the size of abscess was detected by CTE /MRE.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. Patients with CD was diagnosed clinically according to previously established international criteria [9]
3. The diagnosis of stricture, fistula and abdominal abscess was confirmed by ultrasound, CT enterography (CTE), and endoscopy. The bowel stricture should mainly cause by inflammation. Intolerance or failure to steroids or IFX was judged by medical history
4. The disease was in an active period.

Exclusion Criteria:

1. Intolerant to EEN or need emergency surgery
2. The bowel stricture should mainly cause by fibrosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All consecutive adult active CD patients followed up in our center and had been diagnosed with disease complications including stricture, intestinal fistula, abdominal abscess or no response to drugs. Patients were recruited from July 2013 to July 2015.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2013-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Clinical remission after 12 weeks EEN | July 2013 to October 2015
  The Crohn's disease activity index (CDAI)<150 was taken as achieving clinical remission.
Mucosal healing after EEN | July 2013 to October 2015
  Mucosal healing was assessed under endoscopy with SES-CD.

SECONDARY OUTCOMES:
The high sensitivity C-reactive protein (mg/L) -Inflammatory parameter assessment | baseline, week 4 and week 12
  The high sensitivity C-reactive protein (mg/L) was evaluated at baseline, week 4 and week 12.
Inflammatory parameter assessment | baseline, week 4 and week 12
  The platelet (10*9/L) was evaluated at baseline, week 4 and week 12.
The body mass nutritional parameter assessment | baseline, week 4 and week 12
  The body mass was evaluated at baseline, week 4 and week 12.
The albumin (g/L)- nutritional parameter assessment | baseline, week 4 and week 12
  The albumin (g/L) was evaluated at baseline, week 4 and week 12.